CLINICAL TRIAL: NCT00221065
Title: Influence of CPAP on Cognitive Function and Outcome of Stroke Patients With Obstructive Apnea
Brief Title: Effect of Continuous Positive Airway Pressure (CPAP) on Cognitive and Functional Performance in Stroke Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Douglas Bradley, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRI REB 04-043; TRI REB 04-043; NCT00375479 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Sleep Apnea, Obstructive; Cerebrovascular Accident
Keywords: Sleep Apnea Syndromes; Cerebrovascular Accident
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stroke; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Control
- 2 (Experimental): CPAP
  Interventions: Device: Nasal Continuous positive airway pressure - Tyco 420G

INTERVENTIONS:
Device: Nasal Continuous positive airway pressure - Tyco 420G — CPAP at determined pressure nightly for 1 month
  Other Names: Tyco CPAP machines 420 G
  Arms: 2

SUMMARY:
" Obstructive sleep apnea"(OSA) is a sleep breathing disorder. When a person with OSA tries to sleep the back of the throat closes and blocks the flow of air into lungs.When this happens, a person's sleep is disrupted, causing minor awakenings(which the individual may not recognize). This occurs many times throughout the night, causing poor sleep quality,excessive daytime sleepiness, poor concentration, and sometimes depression.It is possible that poor outcomes observed in stroke patients with OSA result from these neurocognitive phenomena, presumably by reducing effective participation in rehabilitation activities.OSA is treated with nasal continuous positive airway pressure(CPAP).CPAP therapy keeps the back of the throat open so that airflow is never blocked.The study is designed to investigate whether treatment of OSA with CPAP improves the results of rehabilitation.

DETAILED DESCRIPTION:
Stroke occurs as a result of ischemic injury to neural tissue, as a result of cardiogenic or artery to artery embolism or intracranial arterial thrombosis. The traditional vascular risk factors, namely hypertension, diabetes mellitus, tobacco smoking, family history and hyperlipidemia as well as atrial fibrillation are major determinants of stroke risk. Obstructive sleep apnea (OSA) has been shown to be a risk factor for hypertension and,although the association is less strong, atherosclerotic heart disease.There is a high prevalence of OSA amongst stroke patients, on the order of 60 to 70%, which is tenfold higher than in the general healthy population. Recently, it has been shown that, in stroke patients undergoing inpatient rehabilitation,the presence of OSA predicts both a poor functional outcome and greater length of hospitalization in the rehabilitation unit, even after adjustment for stroke severity.

We propose to examine the effect of CPAP therapy on the neuropsychological and functional outcomes of stroke patients with OSA admitted to the Toronto Rehabilitation Institute Stroke Rehabilitation Unit in a prospective, randomized study. We hypothesize that, in stroke patients with OSA, CPAP therapy will improve indices of vigilance, attention, and cognitive performances well as motor function(as it does in OSA patients without stroke)when compared to those not treated with CPAP. Furthermore,we hypothesize that the outcome of rehabilitation, as assessed by neuropsychological and motor indices, will be improved in these patients.

ELIGIBILITY:
Inclusion Criteria:

* completed embolic, thrombo-embolic or hemorrhagic subacute strokes admitted within 3 weeks of stroke onset to the SRU of TRI.
* all subjects must be able to follow simple commands in English based upon the Speech Language therapist's intake assessment and have competency to provide informed consent to participate in the study.

Exclusion Criteria:

* brainstem strokes due to increased aspiration risk with CPAP.
* patients with previously diagnosed OSA or stroke.
* diseases primarily or frequently affecting the central nervous system, including dementia, Parkinson's disease, multiple sclerosis,Huntington's disease or Lupus.
* history of a psychotic disorder
* stroke secondary to traumatic brain injury.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Neurological and functional scales | 1 month

SECONDARY OUTCOMES:
Measurements of severity of obstructive sleep apnea and sleep structure | 1 month
Epworth Sleepiness Scale | 1 month
Stanford Sleepiness Scale | 1 month
Participation Assessment Scale | 1 month
Neuropsychological tests(other than primary outcomes) | 1 month
Neurophysiological tests (other than primary outcomes) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Douglas T Bradley, MD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kaneko Y, Floras JS, Usui K, Plante J, Tkacova R, Kubo T, Ando S, Bradley TD. Cardiovascular effects of continuous positive airway pressure in patients with heart failure and obstructive sleep apnea. N Engl J Med. 2003 Mar 27;348(13):1233-41. doi: 10.1056/NEJMoa022479. PMID 12660387
- [Derived] Ryan CM, Bayley M, Green R, Murray BJ, Bradley TD. Influence of continuous positive airway pressure on outcomes of rehabilitation in stroke patients with obstructive sleep apnea. Stroke. 2011 Apr;42(4):1062-7. doi: 10.1161/STROKEAHA.110.597468. Epub 2011 Mar 3. PMID 21372306